CLINICAL TRIAL: NCT00963144
Title: Diagnosis and Response to Treatment Using a Reliable Gerd Questionnaire-an In Clinical Practise Study
Brief Title: Diagnosis and Response to Treatment Using a Reliable Gastroesophageal Reflux Disease (GERD) Questionnaire: An In Clinical Practice Study
Acronym: GQS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-GMY-DUM-2009/1
Record Dates: First submitted 2009-08-12; First posted 2009-08-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gerd Questionnaire
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine the applicability and utility of Gerd Q in the diagnosis of GERD and in the assessment of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender aged between 18-79 years of age
* Patients must be having symptoms of gastroesophageal reflux disease

Exclusion Criteria:

* None

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the applicability and utility of Gerd Q in the diagnosis of GERD and assessment of treatment response | The applicability and utility of the Gerd Questionnaire will be done on 2 vists- Day 1 and Day 30

SECONDARY OUTCOMES:
To assess and monitor the treatment response of patients diagnosed with GERD | The monitoring and assessment of treatment response using the Gerd Questionnaire will be done on 2 vists-Day 1 and Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Goh Khean Lee, MBBS, MRCP, FRCP, Principal Investigator — Faculty of Medicine, University of Malaya Medical Center (UMMC),
Locations (2):
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor